CLINICAL TRIAL: NCT02824016
Title: A Prospective Multicentric Evaluation of the Rate of Incidence of Hypothyroidism After Supraclavicular Irradiation for Breast Cancer
Brief Title: Evaluation of Hypothyroidism Incidence After Breast Cancer Supraclavicular Irradiation
Acronym: EPITHERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jean-Godinot (Other)
Responsible Party: Principal Investigator, Tan Dat NGUYEN, Professor, Institut Jean-Godinot
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2013-A00755-40; 2011-A00822-39 (Other: RCB identifier (ANSM)); 2013-A00755-40 (Other: RCB identifier (ANSM))
Record Dates: First submitted 2014-08-25; First posted 2016-07-06 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Irradiation; Adverse Effect; Irradiation Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with supraclavicular irradiation (Active Comparator): Patients received supraclavicular irradiation according to local policies. Biological samples were obtained in order to evaluate hypothyroidism during the follow-up period
  Interventions: Biological: biological sample; Radiation: supraclavicular irradiation
- without supraclavicular irradiation (Active Comparator): Patients did not receive supraclavicular irradiation according to local policies. Biological samples were obtained in order to evaluate hypothyroidism during the follow-up period
  Interventions: Biological: biological sample

INTERVENTIONS:
Biological: biological sample — T4, thyrotropic-stimulating hormone (TSH) and Thyroglobulin antibody were systematically measured
Radiation: supraclavicular irradiation — Irradiation of the homolateral supraclavicular area delivering 46 Gy in 23 fractions
  Arms: with supraclavicular irradiation

SUMMARY:
Prospective, multicentric, comparative, non randomised, in current care.

Primary objective:

* To evaluate the incidence of hypothyroidism in breast cancer patients treated by radiotherapy including the supra-clavicular area over a period of 5 years (60 months).

Secondary objectives :

* To calculate the dose of irradiation received by thyroid gland during the treatment.
* To compare the rate of incidence of hypothyroidism in women who received a supra-clavicular irradiation (group 1)and in those who did not (group 2).
* To estimate and compare the rate of incidence of chronic thyroid lesions in the 2 groups.
* To look for predictive factors of hypothyroidism de novo in group 1 women particularly regarding the dose-volume parameters.
* To propose recommendations for the thyroid follow-up after supra-clavicular irradiation.

DETAILED DESCRIPTION:
Prospective, multicentric, comparative, non randomised, in current care study

2 patient groups, non randomised, according to the necessity or not to perform a supra-clavicular irradiation:

* Group 1 : patients receiving a supra-clavicular irradiation
* Group 2 : patients not receiving a supra-clavicular irradiation.

Schedule

Projected inclusion duration of 18 months (duration to possibly adapt in order to obtain the number of required patients)

Intermediate study of the results in 30 months

Duration of follow-up of 60 months

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18
* Non metastatic breast cancer, histologically proved, whatever T and N stages and receptors status.
* Breast cancer treated by surgery (either initial treatment then biotherapies and/or neoadjuvant chemotherapy, either secondarily after biotherapies and/or neoadjuvant chemotherapy, either without chemotherapy and/or biotherapies)
* Breast cancer requiring an adjuvant radiotherapy
* Treatment by radiotherapy made in participating centers
* Information of patient and signature of the informed consent.

Exclusion Criteria:

* Pre-existent dysthyroidism revealed before radiotherapy or at inclusion checkup (THS lower or superior to the standard of the laboratory, whatever the rate of free T4)
* History of thyroid surgery
* Bilateral breast cancer
* History of cervical and/or supra-clavicular radiotherapy
* Lack of social security insurance
* Subjects deprived of free behavior or under administrative control

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse effects on thyroid function as assessed by CTCAE v4.0 | Outcome measures will be assessed every 6 months up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Yacine MERROUCHE, MD, Study Director — Institut Jean-Godinot
Locations (3):
- France (3):
  - Institut Jean Godinot, Reims
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided